CLINICAL TRIAL: NCT02460926
Title: Acute Phase Response Following Full Mouth Versus Quadrant Non-Surgical Periodontal Treatment. A Randomized Clinical Trial
Brief Title: Acute Phase Response & Periodontal Treatment
Acronym: PERIOSYST-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Collaborators: Eastman Dental Insitute and Hospital (Other)
Responsible Party: Principal Investigator, Filippo Graziani, DDS MClinDent PhD, Associate Professor, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3399/11
Record Dates: First submitted 2015-05-28; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Periodontal Diseases
Keywords: Scaling and root planning; C-reactive protein
MeSH Terms: conditions — Periodontal Diseases | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scaling & Root Planing - Quadrant (Experimental): Periodontal treatment (PT), consisting in both supra- and sub-gingival mechanical instrumentation of the root surface (scaling and root planing), was performed by a single periodontist . Treatment was provided using both hand and ultrasonic instrumentation with fine tips. Local anaesthesia was used when needed and no time constraints were enforced. Q-SRP patients received four quadrants sessions of PT with an interval of 1 week between sessions
  Interventions: Procedure: Scaling & Root Planing
- Scaling & Root Planing - Full Mouth (Experimental): Periodontal treatment (PT), consisting in both supra- and sub-gingival mechanical instrumentation of the root surface (scaling and root planing), was performed by a single periodontist . Treatment was provided using both hand and ultrasonic instrumentation with fine tips. Local anaesthesia was used when needed and no time constraints were enforced. FM-SRP patients received treatment within 24 hrs in two separate sessions, one side of the mouth for each session: two quadrants were instrumented in an afternoon session, whereas the other two were instrumented the following morning
  Interventions: Procedure: Scaling & Root Planing

INTERVENTIONS:
Procedure: Scaling & Root Planing — It consists in the non-surgical debridement of the sub gingival area affected by periodontal disease
  Other Names: SRP

SUMMARY:
This study has compared quadrant scaling and root planing (Q-SRP) versus intensive treatment performed within 24 hours (FM-SRP) in terms of acute phase responses following treatment of periodontal disease. The primary aim was to compare the differences in CRP acute increase following FM-SRP versus Q-SRP therapy (24 hours after therapy). Secondary outcomes included changes in a broad array of inflammatory and endothelial injury markers between groups. Patients were randomly assigned to either FM-SRP and Q-SRP. Data indicated that non-surgical periodontal therapy performed within 24 hours induced greater perturbations of systemic inflammation compared to conventional treatment.

DETAILED DESCRIPTION:
Aim. A moderate acute-phase response occurs 24 hours following full-mouth non-surgical treatment (FM-SRP). Aim of this study will be to compare quadrant scaling (Q-SRP) versus FM-SRP in terms of systemic acute (24 hours) and medium-term (3 months) inflammation.

Material & Methods. 38 periodontitis-affected subjects will be randomly allocated to FM-SRP or Q-SRP after a baseline visit. Periodontal and anthropometric parameters, such as systolic and diastolic bood pressure, BMI and temperature, will be collected at baseline and 3 months. Serum samples will be drawn at baseline, 1, 7 and 90 days after treatment. High sensitivity assays for a broad array of inflammatory (PCR, IL-6, TNF-alpha) and endothelial assays will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with probing pocket depths (PPD) ≥5 mm,
* bleeding on probing on at least 25% of their total sites
* documented radiographic alveolar bone loss

Exclusion Criteria:

* age earlier than 18 and older than 70 years;
* pregnant or lactating females;
* females using contraceptive methods;
* reported diagnosis of any systemic illnesses including cardiovascular, renal and liver diseases;
* any pharmacological treatment within the 3 months before the beginning of the study;
* PT in the previous 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
C reactive Protein | 24 Hours

SECONDARY OUTCOMES:
C reactive Protein | 7 days, 90 days
Tumor Necrosis Factor - alpha | 24 Hours, 7 days, 90 days
Interleukin - 6 | 24 Hours, 7 days, 90 days
periodontal pocket depth (PPD) | 90 days
  mean in mm
periodontal pocket depth (PPD) | 90 days
  mean in site > 4mm
clinical attachment level (CAL) | 90 days
  mean in mm
number of pockets > 4 mm | 90 days
  number of pockets > 4 mm
Full Mouth Plaque Score | 90 days
  presence/absence of dental plaque in percentual values
Full Mouth Bleeding Score | 90 days
  presence/absence of sites bleeding on probing in percentual values

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Graziani, DDS, PhD, Principal Investigator — University of Pisa

REFERENCES:
- [Background] Graziani F, Cei S, La Ferla F, Vano M, Gabriele M, Tonetti M. Effects of non-surgical periodontal therapy on the glomerular filtration rate of the kidney: an exploratory trial. J Clin Periodontol. 2010 Jul;37(7):638-43. doi: 10.1111/j.1600-051X.2010.01578.x. Epub 2010 May 25. PMID 20500539
- [Result] Graziani F, Cei S, Tonetti M, Paolantonio M, Serio R, Sammartino G, Gabriele M, D'Aiuto F. Systemic inflammation following non-surgical and surgical periodontal therapy. J Clin Periodontol. 2010 Sep;37(9):848-54. doi: 10.1111/j.1600-051X.2010.01585.x. Epub 2010 Jun 4. PMID 20546085